CLINICAL TRIAL: NCT01313624
Title: A Phase 3, Double-Blind, Multicenter, Randomized, Placebo-Controlled Trial Evaluating Repeated Courses of Aztreonam for Inhalation Solution in Subjects With Non-CF Bronchiectasis and Gram-Negative Endobronchial Infection
Brief Title: Safety and Effectiveness of AZLI (an Inhaled Antibiotic) in Adults With Non-Cystic Fibrosis Bronchiectasis
Acronym: AIR-BX1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-219-0101
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZLI-AZLI (Experimental): Participants were randomized to receive blinded AZLI for 2 cycles of 28 days on treatment with each cycle followed by 28 days off treatment, followed by open-label AZLI for 28 days plus 56 days of treatment-free follow-up.
  Interventions: Drug: AZLI
- Placebo-AZLI (Placebo Comparator): Participants were randomized to receive blinded placebo to match AZLI for 2 cycles of 28 days on treatment with each cycle followed by 28 days off treatment, followed by open-label AZLI for 28 days plus 56 days of treatment-free follow-up.
  Interventions: Drug: AZLI; Drug: Placebo

INTERVENTIONS:
Drug: AZLI — AZLI 75 mg reconstituted with diluent and administered via nebulizer three times daily
Drug: Placebo — Placebo to match AZLI administered via nebulizer three times daily
  Arms: Placebo-AZLI

SUMMARY:
The AIR-BX1 study enrolled people with non-cystic fibrosis (non-CF) bronchiectasis and gram-negative airway infection. Participants received two 28-day courses of either Aztreonam for Inhalation Solution (AZLI) or placebo taken 3 times a day. Each course was followed by a 28-day off-drug period. Following the two blinded courses, all participants received a 28-day course of open-label AZLI then were followed for an additional 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female 18 years or older with non-CF bronchiectasis
* Chronic sputum production on most days
* Positive sputum culture for gram-negative organisms
* Must have met lung function requirements

Exclusion Criteria:

* History of CF
* Hospitalized within 14 days prior to joining the study
* Previous exposure to AZLI
* Pregnant, breastfeeding, or unwilling to follow contraceptive measures for the study
* Must have met liver and kidney function requirements
* Continuous oxygen use of greater than 2 liters per minute (supplemental oxygen with activity and at night was allowed)
* Treatment for nontuberculous mycobacteria infection or active mycobacterium tuberculosis infection within 1 year of enrollment
* Other serious medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Barker, MD, Principal Investigator — Oregon Health and Science University
Locations (60):
- United States (36):
  - Pulmonary Associates, Phoenix, Arizona
  - Arizona Pulmonary Specialists, LTD, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center Heart and Lung Institute, Phoenix, Arizona
  - Arizona Pulmonary Specialists, Scottsdale, Arizona
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - UC Davis Medical Center Division of Pulmonary, Critical Care and Sleep Medicine, Sacramento, California
  - Landon Pediatric Foundation, Ventura, California
  - National Jewish Health, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Bay Area Chest Physicians, Clearwater, Florida
  - University of Florida, Gainesville, Florida
  - Pulmonary Disease Specialists (PDS) Research, Kissimmee, Florida
  - University of Miami - Miller School of Medicine, Miami, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Atlanta Pulmonary Group, Atlanta, Georgia
  - Pulmonary and Critical Care Associates of Baltimore, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Cardio Pulmonary Research at St. Luke's Hospital, Chesterfield, Missouri
  - Albany Medical Center, Albany, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Winthrop University Hospital - Clinical Trials Center, Mineola, New York
  - St. Luke's Roosevelt Hospital, New York, New York
  - University of Cincinnati / UC Health, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania Medical Center - Pulmonary, Allergy & Critical Care Division, Philadelphia, Pennsylvania
  - Asthma Allergy & Pulmonary Associates, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Metroplex Pulmonary and Sleep Center, McKinney, Texas
  - Alamo Clinical Research Associates, San Antonio, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas
  - University of Virginia Pulmonary and Critical Care, Charlottesville, Virginia
  - Inova Fairfax Hospital/ Heart and Vascular Institute Advanced Lung Disease and Transplant Center, Falls Church, Virginia
  - Swedish Medical Center/Minor James Clinic, Seattle, Washington
  - Multicare Pulmonary Specialist, Tacoma, Washington
- Australia (15):
  - Concord Hospital, Concord, New South Wales
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Woolcock Institute of Medical Research, Glebe, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Royal Perth Hospital, Perth, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Mater Adult Hospital, Brisbane, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Royla Adelaide Hospital, Adelaide, South Australia
  - Repatriation General Hospital, Daws Park, South Australia
  - Respiratory Clinical Trials, Toorak Gardens, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Peninsula Health, Frankston, Victoria
  - Alfred Hospital, Westmead, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Canada (9):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Kelowna Respiratory and Allergy Clinic, Kelowna, British Columbia
  - The Lung Centre at Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital Pacific Lung Research, Vancouver, British Columbia
  - Kingston General Hospital / Queen's University, Kingston, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Dr. Anil Dhar Private Practice, Windsor, Ontario
  - Centre Hospitalier de L'Université de Montréal Hotel Dieu, Montreal, Quebec

REFERENCES:
- [Derived] Barker AF, O'Donnell AE, Flume P, Thompson PJ, Ruzi JD, de Gracia J, Boersma WG, De Soyza A, Shao L, Zhang J, Haas L, Lewis SA, Leitzinger S, Montgomery AB, McKevitt MT, Gossage D, Quittner AL, O'Riordan TG. Aztreonam for inhalation solution in patients with non-cystic fibrosis bronchiectasis (AIR-BX1 and AIR-BX2): two randomised double-blind, placebo-controlled phase 3 trials. Lancet Respir Med. 2014 Sep;2(9):738-49. doi: 10.1016/S2213-2600(14)70165-1. Epub 2014 Aug 18. PMID 25154045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in a total of 57 study sites in the United States, Canada, and Australia. The first participant was screened on 25 April 2011. The last participant observation was on 04 June 2013.
Pre-assignment Details: 348 participants were screened and 266 were randomized and treated, and comprise the Safety Analysis Set and the Intent-to-Treat (ITT) Analysis Set.
Groups:
- AZLI-AZLI: Participants were randomized to receive blinded Aztreonam for Inhalation Solution (AZLI) 75 mg three times daily via investigational nebulizer for 2 cycles of 28 days on treatment with each cycle followed by 28 days off treatment, followed by open-label AZLI 75 mg three times daily for 28 days plus 56 days of treatment-free follow-up.
- Placebo-AZLI: Participants were randomized to receive blinded placebo to match AZLI three times daily via investigational nebulizer for 2 cycles of 28 days on treatment with each cycle followed by 28 days off treatment, followed by open-label AZLI 75 mg three times daily for 28 days plus 56 days of treatment-free follow-up.
Period: Double-Blind Phase
Arm/Group | AZLI-AZLI | Placebo-AZLI
Started | 134 | 132
Completed | 96 | 122
Not Completed | 38 | 10
Not completed — Adverse Event | 27 | 4
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Period: Open-Label Phase
Arm/Group | AZLI-AZLI | Placebo-AZLI
Started | 96 | 122
Completed | 92 | 109
Not Completed | 4 | 13
Not completed — Adverse Event | 1 | 10
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: ITT Analysis Set
Groups:
- AZLI-AZLI: Participants were randomized to receive blinded AZLI 75 mg three times daily via investigational nebulizer for 2 cycles of 28 days on treatment with each cycle followed by 28 days off treatment, followed by open-label AZLI 75 mg three times daily for 28 days plus 56 days of treatment-free follow-up.
- Placebo-AZLI: Participants were randomized to receive blinded placebo to match AZLI three times daily via investigational nebulizer for 2 cycles of 28 days on treatment with each cycle each followed by 28 days off treatment, followed by open-label AZLI 75 mg three times daily for 28 days plus 56 days of treatment-free follow-up.
- Total: Total of all reporting groups
Arm/Group | AZLI-AZLI | Placebo-AZLI | Total
Number analyzed (Participants) | 134 | 132 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (12.92) | 64.9 (12.11) | 64.6 (12.51)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 54 | 107
  >=65 years | 81 | 78 | 159
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 97 | 181
  Male | 50 | 35 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 23
  Not Hispanic or Latino | 121 | 121 | 242
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 121 | 119 | 240
  African-American | 3 | 6 | 9
  Asian | 5 | 3 | 8
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 4 | 3 | 7
  Not Permitted | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 86 | 79 | 165
  Canada | 17 | 11 | 28
  Australia | 31 | 42 | 73
QOL-B Respiratory Symptom Score [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life Questionnaire-Bronchiectasis (QOL-B) overall score was scaled from 0-100 with higher scores representing better quality of life.
  units on a scale | 55.0 (19.32) | 55.5 (19.26) | 55.2 (19.26)

OUTCOME MEASURES:

1. Primary Outcome: Change in QOL-B Respiratory Symptoms Score at Day 28
Description: The mean (SD) change in the Respiratory Symptoms score on the Quality of Life Questionnaire-Bronchiectasis (QOL-B) was measured from baseline to the end of Course 1 (Day 28). The QOL-B respiratory symptoms score was transformed onto a scale of 0-100, with higher scores representing a better quality of life.
Time Frame: Baseline to Day 28
Population: Participants in the ITT Analysis Set with scores at both baseline and Day 28 were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AZLI-AZLI | Placebo-AZLI
Number analyzed (Participants) | 117 | 124
units on a scale | 7.4 (21.37) | 5.7 (13.62)
Statistical Analysis 1: Comparison: AZLI-AZLI vs Placebo-AZLI; Test type: Superiority or Other; p = 0.68, MMRM — P-value was based on T-test from mixed-effect model repeated measures (MMRM); Difference in least squares mean = 0.8, 95% CI 2-sided [-3.1 to 4.7]

2. Secondary Outcome: Change in QOL-B Respiratory Symptoms Score at Day 84
Description: The mean (SD) change in the Respiratory Symptoms score on the QOL-B was measured from baseline to the end of Course 2 (Day 84). The QOL-B respiratory symptoms score was transformed onto a scale of 0-100, with higher scores representing a better quality of life.
Time Frame: Baseline to Day 84
Population: Participants in the ITT Analysis Set with scores at both baseline and Day 84 were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AZLI-AZLI | Placebo-AZLI
Number analyzed (Participants) | 108 | 122
units on a scale | 7.4 (21.67) | 4.7 (17.24)
Statistical Analysis 1: Comparison: AZLI-AZLI vs Placebo-AZLI; Test type: Superiority or Other; p = 0.56, MMRM — P-value was based on T-test from mixed-effect model repeated measures (MMRM); Difference in least squares mean = 1.3, 95% CI 2-sided [-3.0 to 5.6]

3. Secondary Outcome: Time to Protocol-Defined Exacerbation (PDE)
Description: Protocol-defined exacerbation was defined as an acute worsening of respiratory disease that triggered the initiation of a non-study antibiotic meeting at least 3 major criteria, or 2 major and at least 2 minor criteria.
  * Major Criteria: increased sputum production; increased discoloration of sputum; increased dyspnea; increased cough
  * Minor Criteria: fever (> 38º C) measured during clinic visit; increased malaise or fatigue; forced expiratory volume in 1 second (FEV1) (L) or forced vital capacity (FVC) decreased > 10% from baseline; new or increased hemoptysis
Time Frame: Baseline to Day 112
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | AZLI-AZLI | Placebo-AZLI
Number analyzed (Participants) | 134 | 132
days | NA [NA to NA] — At least 50% of participants must have had a PDE in order to compute the median days to PDE. Fewer than 50% of participants in this group had a PDE, so median days to PDE could not be computed. | 120 [117.0 to NA] — The 95% upper confidence interval (CI) could not be estimated due to an insufficient number of PDE events.

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after the last dose of study drug.
Groups:
- AZLI-AZLI (Double-Blind): Adverse events for this reporting group were reported from baseline to Day 112 while participants were receiving double-blind AZLI; participants were randomized to receive blinded placebo to match AZLI three times daily via investigational nebulizer for 2 cycles of 28 days on treatment with each cycle followed by 28 days off treatment, followed by open-label AZLI 75 mg three times daily for 28 days plus 56 days of treatment-free follow-up.
- Placebo-AZLI (Double-Blind): Adverse events for this reporting group were reported from baseline to Day 112 while participants were receiving double-blind placebo; participants were randomized to receive blinded placebo to match AZLI three times daily via investigational nebulizer for 2 cycles of 28 days on treatment with each cycle followed by 28 days off treatment, followed by open-label AZLI 75 mg three times daily for 28 days plus 56 days of treatment-free follow-up.
- AZLI-AZLI (Open-Label); Placebo-AZLI (Open-Label): Adverse events for this reporting group were reported from Day 112 to Day 196 plus 30 days while participants were receiving open-label AZLI; participants were randomized to receive blinded placebo to match AZLI three times daily via investigational nebulizer for 2 cycles of 28 days on treatment with each cycle followed by 28 days off treatment, followed by open-label AZLI 75 mg three times daily for 28 days plus 56 days of treatment-free follow-up.
Arm/Group | AZLI-AZLI (Double-Blind) | Placebo-AZLI (Double-Blind) | AZLI-AZLI (Open-Label) | Placebo-AZLI (Open-Label)
Serious Adverse Events (participants affected / at risk) | 28/134 | 13/132 | 9/96 | 18/122
Other Adverse Events (participants affected / at risk) | 116/134 | 102/132 | 54/96 | 76/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI-AZLI (Double-Blind) (N=134) | Placebo-AZLI (Double-Blind) (N=132) | AZLI-AZLI (Open-Label) (N=96) | Placebo-AZLI (Open-Label) (N=122)
Infective exacerbation of bronchiectasis (Infections and infestations) | 5 | 4 | 5 | 7
Pneumonia (Infections and infestations) | 5 | 1 | 2 | 6
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Orthostatic intolerance (Nervous system disorders) | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 2
Type IV hypersensitivity reaction (Immune system disorders) | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI-AZLI (Double-Blind) (N=134) | Placebo-AZLI (Double-Blind) (N=132) | AZLI-AZLI (Open-Label) (N=96) | Placebo-AZLI (Open-Label) (N=122)
Cough (Respiratory, thoracic and mediastinal disorders) | 69 | 57 | 35 | 50
Sputum Increased (Respiratory, thoracic and mediastinal disorders) | 62 | 48 | 29 | 36
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 42 | 33 | 24 | 26
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 | 12 | 5 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 73 | 47 | 31 | 47
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 17 | 4 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 21 | 14 | 6 | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 14 | 3 | 6 | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 0 | 0
Fatigue (General disorders) | 56 | 29 | 22 | 19
Malaise (General disorders) | 11 | 14 | 5 | 5
Pyrexia (General disorders) | 32 | 16 | 7 | 12
Non-cardiac chest pain (General disorders) | 20 | 14 | 6 | 8
Chills (General disorders) | 18 | 6 | 6 | 3
Oedema peripheral (General disorders) | 7 | 6 | 0 | 0
Headache (Nervous system disorders) | 21 | 23 | 5 | 7
Sinus headache (Nervous system disorders) | 8 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 10 | 6 | 0 | 0
Nausea (Gastrointestinal disorders) | 13 | 11 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 6 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 12 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 5 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years